CLINICAL TRIAL: NCT00245011
Title: High Dose Samarium-153 With Peripheral Blood Stem Cell Support in High Risk Osteogenic Sarcoma
Brief Title: Samarium Sm 153 and Stem Cell Transplant Followed By Radiation Therapy Patients With Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0347; JHOC-J0347 (Other: Johns Hopkins University Clinical Research Office (CRO)); 03-09-08-02 (Other: JHM IRB); CDR0000447134 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Sarcoma
Keywords: recurrent osteosarcoma; metastatic osteosarcoma; localized osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — Filgrastim; Ifosfamide; Peripheral Blood Stem Cell Transplantation; samarium Sm-153 lexidronam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Samarium-153 (Experimental): Cytoxan+Ifosfamide, Filgrastim pre samarium.'Sm-EDTMP (low dose). once counts recover, Sm-EDTMP (high dose) given. Peripheral blood stem cell transplantation is done 14 days later.
  Interventions: Biological: filgrastim; Drug: ifosfamide; Procedure: peripheral blood stem cell transplantation; Radiation: Sm-EDTMP (low dose); Radiation: sm-EDTMP (higher dose)

INTERVENTIONS:
Biological: filgrastim — Filgrastim will be administered post post chemotherapy until target WBC (white blood cell) count is achieved.
  Other Names: Neupogen
Drug: ifosfamide — Ifosfamide administered IV.
  Other Names: Ifex
Procedure: peripheral blood stem cell transplantation — Peripheral blood stem cell transplantation is done 14 days after 2nd dose of Samarium is delivered
Radiation: Sm-EDTMP (low dose) — Sm-EDTMP (low dose) administered after autologous stem cell collection
Radiation: sm-EDTMP (higher dose) — Upon blood cell count recovery from Sm-EDTMP (low dose), Sm-EDTMP (higher dose) is administered followed in 14 days by peripheral blood stem cell transplantation.

SUMMARY:
RATIONALE: Radioactive drugs, such as samarium Sm 153 lexidronam pentasodium, may carry radiation directly to tumor cells and not harm normal cells. A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy and samarium Sm 153 lexidronam pentasodium. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving samarium Sm 153 lexidronam pentasodium together with a peripheral stem cell transplant and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving samarium Sm 153 lexidronam pentasodium together with autologous stem cell transplant and radiation therapy works in treating patients with recurrent or refractory, metastatic, or unresectable osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response in patients with recurrent or refractory, metastatic, or unresectable osteosarcoma treated with high-dose samarium Sm 153 lexidronam pentasodium (^153Sm-EDTMP) and autologous peripheral blood stem cell transplantation followed by external-beam radiotherapy.
* Correlate the amount of radiation delivered to a tumor with low-dose ^153Sm-EDTMP with that of high-dose ^153Sm-EDTMP in patients treated with this regimen.

Secondary

* Determine the overall and progression-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the long-term effects of this regimen in these patients.
* Determine the predictive value of fludeoxyglucose F 18 positron emission tomography (FDG-PET), diffusion-weighted MRI, and magnetic resonance spectroscopy for evaluation of treatment response in patients treated with this regimen.

OUTLINE: Patients are stratified according to resectability of the primary tumor (recurrent, refractory, or very high-risk disease vs unresectable primary tumor).

* Mobilization and collection of autologous peripheral blood stem cells (PBSCs)* : Patients receive ifosfamide IV daily for 5 days followed by filgrastim (G-CSF) subcutaneously daily. Patients then undergo leukapheresis for collection of autologous PBSCs until ≥ 2 x 10^6 CD34 (cluster of differentiation 34)-positive cells/kg are collected.

NOTE: *Patients who have undergone PBSC collection before study entry proceed to high-dose samarium Sm 153 lexidronam pentasodium (153Sm-EDTMP) infusion without mobilization and collection of autologous PBSCs.

* 153Sm-EDTMP infusion: Patients receive a trace dose of ^153Sm-EDTMP** IV over 1-2 minutes and undergo bone scan 4, 24, and 48-72 hours later. Six weeks later, patients receive high-dose ^153Sm-EDTMP IV over 1-2 minutes and undergo repeat bone scans 4, 24, and 48-72 hours later.

NOTE: **Patients may receive the trace dose on protocol JHOC (Johns Hopkins Oncology Center)-J0094.

* Autologous peripheral blood stem cell transplantation (PBSCT): Between 12-14 days after administration of high-dose ^153Sm-EDTMP, patients undergo autologous PBSCT. Beginning 2 days later, patients receive G-CSF IV daily.
* External-beam radiotherapy: Patients then undergo external-beam radiotherapy to the sites of bulky disease.
* Surgery: Some patients may also undergo surgical resection of residual disease. After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
Inclusion

* Diagnosis of osteosarcoma

  * High-risk disease, meeting 1 of the following criteria:

    * Recurrent disease
    * Refractory to conventional therapy
    * Newly diagnosed metastatic disease with ≥ 4 pulmonary nodules or multiple bone lesions
    * Unresectable primary tumor
  * Prior intralesional resection allowed
* Measurable disease by technetium Tc 99m diphosphonate bone scan
* Refractory to all standard therapies or highly unlikely to respond to conventional treatment
* Performance status Karnofsky 60-100%
* Life expectancy more than 8 weeks
* Absolute neutrophil count > 500/mm^3
* Platelet count > 50,000/mm^3
* Creatinine clearance > 70 mL/min OR * Radioisotope glomerular filtration rate normal
* Recovered from prior chemotherapy

Exclusion

* Pregnant or nursing
* Positive pregnancy test for females of childbearing potential
* Fertile patients do not agree to use effective contraception
* Prior radiotherapy to the site of currently active disease
* Concurrent enrollment on protocol JHOC-J0094 allowed

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2004-10; Primary Completion 2008-10 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Loeb, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Senthamizhchelvan S, Hobbs RF, Song H, Frey EC, Zhang Z, Armour E, Wahl RL, Loeb DM, Sgouros G. Tumor dosimetry and response for 153Sm-ethylenediamine tetramethylene phosphonic acid therapy of high-risk osteosarcoma. J Nucl Med. 2012 Feb;53(2):215-24. doi: 10.2967/jnumed.111.096677. Epub 2012 Jan 17. PMID 22251554
- [Result] Loeb DM, Hobbs RF, Okoli A, Chen AR, Cho S, Srinivasan S, Sgouros G, Shokek O, Wharam MD Jr, Scott T, Schwartz CL. Tandem dosing of samarium-153 ethylenediamine tetramethylene phosphoric acid with stem cell support for patients with high-risk osteosarcoma. Cancer. 2010 Dec 1;116(23):5470-8. doi: 10.1002/cncr.25518. Epub 2010 Aug 16. PMID 20715156
- [Result] Loeb DM, Garrett-Mayer E, Hobbs RF, Prideaux AR, Sgouros G, Shokek O, Wharam MD Jr, Scott T, Schwartz CL. Dose-finding study of 153Sm-EDTMP in patients with poor-prognosis osteosarcoma. Cancer. 2009 Jun 1;115(11):2514-22. doi: 10.1002/cncr.24286. PMID 19338063

RESULTS

PARTICIPANT FLOW:
Groups:
- Samarium-153/Stem Cell Transplant/Radiation: Samarium Sm153 Lexidronam Pentasodium (Samarium)/Stem Cell Transplant/Radiation arm: receive Ifosphamide IV in preparation for peripheral blood stem cell transplant followed by collection of stem cells. Samarium is administered after collection of peripheral blood stem cells (PBCT). Once counts recover, while receiving filgrastim daily, a second, higher dose of Samarium-153 is given, followed in 14 days by infusion of the stem cells.
  Filgrastim: administered daily until count recovery Ifosfamide: administered as part of Stem Cell transplant preparation. PBCT: Before administration of Samarium, collection of autologous hematopoietic stem cells Radiation: Radiation Dosimetry performed at 4, 24, 48, and 72 after each infusion of Sm-EDTMP.
  Samarium: First dose is administered after autologous stem cell collection. Second, higher dose, of SM-EDTMP administered after count recover. 14 days after administration of higher dose, patient undergoes autologous stem cell infusion.
Period: Overall Study
Arm/Group | Samarium-153/Stem Cell Transplant/Radiation
Started | 11
Completed | 10 (Subject had disease progression prior to completing study.)
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- Samarium-153/Stem Cell Transplant/Radiation: Samarium Sm153 Lexidronam Pentasodium/Stem Cell Transplant/Radiation arm will receive Ifosphamide IV in preparation for peripheral blood stem cell transplant followed by stem cell collection. Samarium Sm153 Lexidronam Pentasodium is administered after collection of peripheral blood stem cells. Once counts recover, while receiving filgrastim daily, a 2nd, higher dose of Samarium-153 is given, followed in 14 days by stem cell infusion.
  Filgrastim: Filgrastim will be administered every day til count recovery Ifosfamide: Ifosfamide will be administered as part of Stem Cell transplant prep.
  Peripheral blood stem cell transplantation: Before administration of Samarium, collection of autologous hematopoietic stem cells Radiation: Radiation Dosimetry performed at 4, 24, 48, and 72 after each infusion of Sm-EDTMP.
  Samarium Sm 153 lexidronam pentasodium: First dose of Sm-EDTMP administered after autologous stem cell collection. Second, higher dose, of SM-EDTMP administered 7 days later.
Arm/Group | Samarium-153/Stem Cell Transplant/Radiation
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 18 [14 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: WHO (World Health Organization) tumor measurement criteria used to determine response.
Time Frame: 1 week after study treatment
Population: 11 subjects, heavily treated with chemotherapy with osteosarcoma metastatic to bone were enrolled; 10 evaluable for response.
Measure: Number; unit: participants
Groups:
- Samarium-153/Stem Cell Transplant/Radiation: Samarium Sm153 Lexidronam Pentasodium (^153Sm-EDTMP)/Stem Cell Transplant/Radiation arm will receive Ifosphamide IV in preparation for peripheral blood stem cell transplant followed by stem cell harvest. ^153Sm-EDTMP is administered after collection of peripheral blood stem cells. Once counts recover, while receiving filgrastim daily, a 2nd, higher dose of ^153Sm-EDTMP is given, followed in 14 days by stem cell infusion.
  filgrastim: Filgrastim is administered every day til count recovery.
  ifosfamide: Ifosfamide is administered as part of Stem Cell transplant prep.
  peripheral blood stem cell harvesting: completed before administration of ^153Sm-EDTMP, collection of autologous hematopoietic stem cells.
  radiation: Radiation Dosimetry performed at 4, 24, 48, and 72 after each infusion of ^153Sm-EDTMP.
  ^153Sm-EDTMP: First dose is administered after autologous stem cell collection. Second, higher dose, is administered 1 week later.
Arm/Group | Samarium-153/Stem Cell Transplant/Radiation
Number analyzed (Participants) | 10
participants | 10

2. Secondary Outcome: Predictive Value of Imaging Studies
Time Frame: At Time of Tumor Resection
Population: The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and is not available to be reported.
Arm/Group | Samarium-153/Stem Cell Transplant/Radiation
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall and Progression-free Survival After Study Treatment
Time Frame: up to 4 years
Measure: Median (Full Range); unit: days
Arm/Group | Samarium-153/Stem Cell Transplant/Radiation
Number analyzed (Participants) | 11
days
  Overall Survival | NA [NA to NA] — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and is not available to be reported
  Progression-free Survival | 79 [NA to NA] — The PI has left the institution and the only access to the data is from publications. The access to this specific information/data cannot be confirmed and is not available to be reported

4. Secondary Outcome: Toxicity at End of Study Treatment
Time Frame: Continual and at End of Study
Measure: Count of Participants; unit: Participants
Arm/Group | Samarium-153/Stem Cell Transplant/Radiation
Number analyzed (Participants) | 11
Participants
  Delayed numbness and tingling | 3
  Mild hypocalcemia | 1
  Mild - Moderate pancytopenia | 11
  Lymphopenia | 11
  Fever | 5

5. Secondary Outcome: Long Term Side Effects of Infusional Samarium-153 After Study Treatment
Time Frame: Continual
Population: as for outcome 2
Arm/Group | Samarium-153/Stem Cell Transplant/Radiation
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlative Dose of Radiation by Low Dose and High Dose Samarium-153
Time Frame: completion of treatment
Population: as for outcome 2
Arm/Group | Samarium-153/Stem Cell Transplant/Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 weeks; the dose limiting toxicity was defined to be recovery of blood counts by 6 weeks post treatment with SmEDTMP (higher dose). Subjects continued to be monitored until count recovery and indefinitely for survival.
Description: The PI has left the institution and the only access to the data is from publications. The access to all-cause mortality data cannot be confirmed and is not available to be reported.
Groups:
- Samarium-153: Cytoxan+Ifosfamide, Filgrastim pre samarium.'Sm-EDTMP (low dose). once counts recover, Sm-EDTMP (high dose) given. Peripheral blood stem cell transplantation is done 14 days later.
  filgrastim: Filgrastim will be administered post post chemotherapy until target WBC count is achieved.
  ifosfamide: Ifosfamide administered IV.
  peripheral blood stem cell transplantation: Peripheral blood stem cell transplantation is done 14 days after 2nd dose of Samarium is delivered
  Sm-EDTMP (low dose): Sm-EDTMP (low dose) administered after autologous stem cell collection
  sm-EDTMP (higher dose): Upon blood cell count recovery from Sm-EDTMP (low dose), Sm-EDTMP (higher dose) is administered followed in 14 days by peripheral blood stem cell transplantation.
Arm/Group | Samarium-153
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 10/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Samarium-153 (N=11)
Low Platelets (Blood and lymphatic system disorders) | 8 (8) — Grade 3 or 4
Neutorpenia (Blood and lymphatic system disorders) | 8 (8) — Gr 1-2: 3 subjects Gr 3-4: 5 subjects
Anemia (Blood and lymphatic system disorders) | 10 (10) — Gr 1: 10 subjects
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Gr3 increase in size of pleural effusion (disease related). This subject is not evaluable for hematologic recovery.
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — asymptomatic. Grade 3. Resolved spontaneously.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes